CLINICAL TRIAL: NCT05810038
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rimegepant for Migraine Prevention in Chinese Participants
Brief Title: A Study to Learn About the Safety and Effects of Rimegepant to Prevent Migraine in Chinese Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4951019; BHV3000-319 (Other: Alias Study Number)
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Rimegepent; preventive treatment; migraine.
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DBT Rimegepant/OLE Rimegepant (Experimental): DBT Phase (Weeks 1 through 12): Participants will receive a single oral dose of rimegepant orally disintegrating tablet (ODT) EOD for 12 weeks.
  OLE Phase (Weeks 13 through 24): Participants who continue to meet study entry criteria, will enter the OLE phase and receive a single oral dose of rimegepant ODT EOD for 12 weeks. If participants have a migraine on a day that they are not scheduled to dose with rimegepant, they can take one tablet of rimegepant ODT on that calendar day to treat a migraine (as needed [PRN] dosing).
  Interventions: Drug: Rimegepant
- DBT Placebo/OLE Rimegepant (Placebo Comparator): DBT Phase (Weeks 1 through 12): Participants will receive a single oral dose of placebo matching to rimegepant ODT EOD for 12 weeks.
  OLE Phase (Weeks 13 through 24): Participants who continue to meet study entry criteria, will enter the OLE phase and receive a single oral dose of rimegepant ODT EOD for 12 weeks. If participants have a migraine on a day that they are not scheduled to dose with rimegepant, they can take one tablet of rimegepant ODT on that calendar day to treat a migraine (PRN dosing).
  Interventions: Drug: Rimegepant; Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — Rimegepant
  Other Names: PF-07899801, BHV-3000
Drug: Placebo — matching placebo
  Arms: DBT Placebo/OLE Rimegepant

SUMMARY:
The purpose of this study is to learn about the effects of Rimegepant to help prevent migraine.

This study is seeking for participants who:

* Are male and female of 18 years of age or older.
* Have at least 1 year history of migraine .
* Did not take any medication for migraine before the start of this study. The study will go on for around 30 weeks, including 4 Phases and 11 Visits. Participants who are selected for the study will be randomly assigned to treatment groups. After which, the participants will enter a 12-week Double-blind Treatment (DBT) Phase. After finishing the DBT Phase, some selected participants may enter a 12-week Open-label Extension (OLE) Phase. Participants will come back to the study site at the end of Week 24 for the End of Treatment (EOT) Visit. There will be a follow-up Week 2 Visit around 14 days after the EOT visit.

Participants will be asked to take 1 tablet of study medicine every other calendar day. This need to be followed regardless of whether they have a migraine on that day or not. During the OLE Phase only, if a participant has a migraine on a non-scheduled dosing day, they may take 1 tablet of Rimegepant orally disintegrating tablet (ODT) as acute treatment for their migraine, if needed, with a maximum of 1 tablet of Rimegepant per calendar day. The study team will look at how each participant is doing with the study treatment during the regular visits at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

1.Target Population: Participant has at least 1 year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition, including the following:

1. Age of onset of migraines prior to 50 years of age
2. Migraine attacks, on average, lasting 4 to 72 hours if untreated
3. Per participant report, 4 to18 migraine attacks of moderate or severe intensity per month within the last 3 months prior to the Screening Visit (month is defined as 4 weeks for the purpose of this protocol)
4. 6 or more migraine days during Observation Phase
5. Not more than 18 headache days during the Observation Phase
6. Ability to distinguish migraine attacks from tension/cluster headaches.
7. Participants with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Exclusion Criteria:

1. Participant has a history of basilar migraine or hemiplegic migraine.
2. Participants are excluded if they have had no therapeutic response with > 2 of the 9 medication categories of preventive treatment of migraine after an adequate therapeutic trial in the past 3 years per investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Mean change from the Observation Phase (OP) in the number of migraine days per month over the entire Double Blind Treatment (DBT) Phase | OP (up to 4 weeks) and Weeks 1-12 of the DBT phase
  The change from OP (up to 4 weeks) is calculated as the number of monthly migraine days during the 12 weeks of the DBT phase (Weeks 1 to 12) minus number of monthly migraine days during the OP (up to 4 weeks).

SECONDARY OUTCOMES:
Proportion of participants with >= 50% reduction from the OP in the number of moderate to severe migraine days per month over the entire DBT Phase | OP (up to 4 weeks) and Weeks 1-12 of the DBT phase
  A reduction of at least 50% in the mean number of moderate or severe monthly migraine days was determined if the number of moderate or severe monthly migraine days in the 12 weeks of the DBT (Weeks 1 to 12) is less than or equal to half (50%) of the number of moderate or severe monthly migraine days in the OP (up to 4 weeks).
Mean change from the OP in the number of migraine days per month in the first 4 weeks (Weeks 1 to 4) of the DBT Phase. | OP (up to 4 weeks) and Weeks 1-4 of the DBT phase
  The change from OP (up to 4 weeks) is calculated as the number of monthly migraine days during the first 4 weeks of the DBT phase (Weeks 1 to 4) minus number of monthly migraine days during the OP (up to 4 weeks).
Mean change from the OP in the number of migraine days per month in the last 4 weeks (Weeks 9 to 12) of the DBT Phase. | OP (up to 4 weeks) and Weeks 9-12 of the DBT phase
  The change from OP (up to 4 weeks) is calculated as the number of monthly migraine days during the last 4 weeks of the DBT phase (Weeks 9 to 12) minus number of monthly migraine days during the OP (up to 4 weeks).
Mean change from baseline in the MSQoL v2.1 role function - restrictive domain score at Week 12 of the DBT Phase | OP (up to 4 weeks) and Week 12 of the DBT phase
  The change from baseline was calculated as the MSQoL restrictive role function domain score at Week 12 of the DBT phase minus the MSQoL restrictive role function domain score at baseline.
Number of Participants With Adverse Events (AEs), Serious AEs (SAEs) and AEs Leading to Study Drug Discontinuation during the DBT Phase and OLE Phase. | Weeks 1-12 of the DBT phase, and Weeks 13-24 of the OLE phase
  An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition on-treatment in a patient or clinical investigation participant administered an investigational product and that did not necessarily have a causal relationship with this treatment. An SAE is defined as any event that met any of the following criteria: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received an investigational product; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention.
Percentage of participants With Adverse Events (AEs), Serious AEs (SAEs) and AEs Leading to Study Drug Discontinuation during the DBT Phase and OLE Phase. | Weeks 1-12 of the DBT phase, and Weeks 13-24 of the OLE phase
  An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition on-treatment in a patient or clinical investigation participant administered an investigational product and that did not necessarily have a causal relationship with this treatment. An SAE is defined as any event that met any of the following criteria: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received an investigational product; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention.
Number of participants with AST or ALT elevations > 3x ULN concurrent with total bilirubin elevations > 2x ULN on treatment during the DBT Phase and OLE Phase. | Weeks 1-12 of the DBT phase, and Weeks 13-24 of the OLE phase
  Elevations of AST > 3 x ULN concurrent with TBL > 2 x ULN were defined as elevations on the same collection date.
Percentage of participants with AST or ALT elevations > 3x ULN concurrent with total bilirubin elevations > 2x ULN on treatment during the DBT Phase and OLE Phase. | Weeks 1-12 of the DBT phase, and Weeks 13-24 of the OLE phase
  Elevations of AST > 3 x ULN concurrent with TBL > 2 x ULN were defined as elevations on the same collection date.
Number of participants with hepatic-related AEs on treatment during the DBT Phase and OLE Phase. | Weeks 1-12 of the DBT phase, and Weeks 13-24 of the OLE phase
  Hepatic AEs are defined as all preferred terms under the "Hepatic Disorders" Standardized Medical Dictionary (Version 21.1) for Regulatory Activities Query (SMQ), except those preferred terms in the "Congenital, Familial, Neonatal and Genetic Disorders of the Liver" SMQ.
Percentage of participants with hepatic-related AEs on treatment during the DBT Phase and OLE Phase. | Weeks 1-12 of the DBT phase, and Weeks 13-24 of the OLE phase
  Hepatic AEs are defined as all preferred terms under the "Hepatic Disorders" Standardized Medical Dictionary (Version 21.1) for Regulatory Activities Query (SMQ), except those preferred terms in the "Congenital, Familial, Neonatal and Genetic Disorders of the Liver" SMQ.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- China (49):
  - The Second People's hospital of Hefei, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The fourth people's hospital of chongqing, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The 900th Hospital of Joint Logistics Support Force, PLA, Fuzhou, Fujian
  - Lanzhou university second hospital, Lanzhou, Gansu
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Hebei General Hospital, Shijiazhuang, Hebei
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Wuxi No. 2 People's Hospital, Wuxi, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - General Hospital of Ningxia Medical Hospital, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shaanxi
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng people's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - People's Hospital of Rizhao, Rizhao, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated hospital of Kunming Medical University, Kunming, Yunnan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hosptial of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Chongqing University Three Gorges Hospital, Chongqing
  - Tianjin Union Medical Center, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951019
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-319